CLINICAL TRIAL: NCT06091241
Title: ESPBs vs TAPs for Satisfactory Analgesia Following DIEP Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Tara Notarianni, DO, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00150240
Record Dates: First submitted 2023-07-03; First posted 2023-10-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The principal investigator will be unblinded. The study coordinator will be blinded, unable to access procedure notes and randomization assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Erector Spinae Plane blocks (Other): Erector Spinae Plane blocks
  Interventions: Procedure: Pre-operative Erector Spinae Plane block prior to DIEP surgery
- Group 2: Transversus Abdominis Plane blocks (Other): Transversus Abdominis Plane blocks
  Interventions: Procedure: Pre-operative Transversus Abdominus Plane blocks prior to DIEP surgery

INTERVENTIONS:
Procedure: Pre-operative Erector Spinae Plane block prior to DIEP surgery — After obtaining informed consent to participate in the study, patients will be randomized by a computer 50/50 to either the Erector Spinae Plane group or the Transversus Abdominus Plane group at the time of their surgical clinic visit prior to their scheduled surgery. Then on the morning of surgery, the Erector Spinae Plane group will receive a bilateral ultrasound-guided Erector Spinae Plane peripheral nerve block. During this intervention, 0.25% bupivacaine with dexamethasone will be injected below the fascia of the erector spinae muscle group.
  Other Names: ESPBs
  Arms: Group 1: Erector Spinae Plane blocks
Procedure: Pre-operative Transversus Abdominus Plane blocks prior to DIEP surgery — On the morning of surgery, the patients in the TAPs group will receive a bilateral ultrasound-guided Transversus Abdominus plane peripheral nerve block. During this intervention, 0.25% bupivacaine with dexamethasone will be injected into the transversus abdominus plane above the transversus abdominus muscle.
  Other Names: TAPs
  Arms: Group 2: Transversus Abdominis Plane blocks

SUMMARY:
Breast cancer is the second most common cancer diagnosed in American women . For patients who have undergone surgical mastectomy, autologous breast reconstruction is an alternative option to breast implants. Deep Inferior Epigastric Perforator (DIEP) flaps are the gold standard for autologous breast reconstruction . Effective pain control following surgery is imperative and ultrasound-guided bilateral transversus abdominis plane blocks (TAPs) with the infiltration of local anesthetics, such a bupivacaine are a common regional technique of choice . A newer described technique, bilateral Erector Spinae Plane blocks (ESPBs) (which also are an infiltration of local anesthetic) present as an alternative approach for post-operative analgesia. ESPBs have been proven efficacious in reducing intra- and post-operative opioid requirements, lessening the need for rescue analgesics in other similar surgical procedures.

The hypothesis is that preoperative bilateral ESPBs could provide equivalent pain control as a regional analgesic for patients undergoing DIEP flap surgery when compared to preoperative bilateral TAPs

ELIGIBILITY:
Inclusion Criteria:

* Adult women with breast cancer, ASA 1-3, undergoing DIEP flap surgery

Exclusion Criteria:

* Chronic opioid use contraindications to local anesthetics or regional analgesia Inability to communicate intensity of pain on a numeric analog scale

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | 24 hours post injection
  Scale used to measure pain on scale from 0-10 (0 is 'no pain' and 10 is 'the worst pain imaginable')
Mean Morphine Equivalents | 24 hours post injection
  Amount of opioid pain medications administered and converted to morphine equivalents

SECONDARY OUTCOMES:
Numerical Rating Scale | 12 hours post injection
  Scale used to measure pain on scale from 0-10 (0 is 'no pain' and 10 is 'the worst pain imaginable')
Michigan Body Map | 24 hours post injection
  Map used to show body location of worst site of primary pain
Mean Morphine Equivalents | 48 hours post injection
  Amount of opioid pain medications administered and converted to morphine equivalents
Numerical Rating Scale | 48 hours post injection
  Scale used to measure pain on scale from 0-10 (0 is 'no pain' and 10 is 'the worst pain imaginable')
Numerical Rating Scale | 3 months post-operation
  Scale used to measure pain on scale from 0-10 (0 is 'no pain' and 10 is 'the worst pain imaginable')
Numerical Rating Scale | 6 months post-operation
  Scale used to measure pain on scale from 0-10 (0 is 'no pain' and 10 is 'the worst pain imaginable')

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No